CLINICAL TRIAL: NCT00252291
Title: A Phase III Multicenter Study to Demonstrate the Sensitivity and Specificity of Aridol (Mannitol) Challenge to Predict Bronchial Hyperresponsiveness as Manifested by a Positive Exercise Challenge in Subjects Presenting With Signs and Symptoms Suggestive of Asthma But Without a Definitive Diagnosis
Brief Title: Ability of Aridol to Detect Bronchial Hyperresponsiveness in Suspected Asthmatics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Syntara (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: DPM-A-305
Record Dates: First submitted 2005-11-10; First posted 2005-11-11 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Asthma
Keywords: bronchial; hyperresponsiveness
MeSH Terms: conditions — Asthma | interventions — Mannitol; Methacholine Chloride

INTERVENTIONS:
Drug: Aridol
Drug: Methacholine
Procedure: Exercise challenge

SUMMARY:
This is a Phase 3 study to determine the sensitivity and specificity of the Aridol bronchial challenge test to detect bronchial hyperresponsiveness in patients with suspected asthma. Patients with suspected asthma of either gender, aged between 6 and 50 years, with only mildly impaired lung function (FEV1 >70%) are to be tested with three different bronchial hyperresponsiveness challenges (Aridol, exercise and methacholine), and the results compared. A clinical diagnosis will also be made at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Have given informed consent to participate in this study in accordance with local regulations prior to any procedures being performed
2. Have signs and symptoms suggestive of asthma according to the NIH Questionnaire but has not been given a firm diagnosis of asthma or a firm exclusion of the diagnosis of asthma (e.g. has an equivocal diagnosis of asthma or been referred for further investigation of asthma type symptoms)
3. Have at least Step 1 symptoms according to the NAEPPII asthma severity grading
4. Have an FEV1 ≥ 70% of the predicted value at Screening Visit (Visit 1) baseline
5. Be between 6 and 50 years
6. Be able to perform all of the techniques necessary to measure lung function including an exercise challenge, Aridol challenge and methacholine challenge
7. Be able to understand the requirements of the study and be able to complete all of the forms necessary including the NIH Questionnaire
8. Be taking effective birth control if female of childbearing potential

Exclusion Criteria:

1. Use medications six weeks prior to the Screening Visit (Visit 1) or during the study that would interfere with bronchial provocation challenge testing (see Table 1, section 3.3.3.4)
2. Currently use cholinesterase-inhibitor medication (for myasthenia gravis)
3. Have had upper or lower respiratory tract infection within the previous 4 weeks
4. Have known aortic or cerebral aneurysm, cirrhosis or portal hypertension
5. Have had recent major surgery
6. Have had recent cataract surgery
7. Have a history of heart disease that would increase risk of performing exercise, methacholine or Aridol challenge
8. Have had cardiac ischemia or malignant arrhythmias
9. Have uncontrolled hypertension (systolic blood pressure ≥ 180 and diastolic blood pressure ≥ 100)
10. Have orthopedic limitations
11. Have smoked within the past year (average > 1 cigarette per week), or have a ≥ 10 pack year smoking history
12. Have other chronic restrictive or obstructive pulmonary diseases (cystic fibrosis, COPD, bronchiectasis, chronic bronchitis, emphysema, tuberculosis, pulmonary carcinoma, pulmonary fibrosis, pulmonary hypertension, hypercapnia)
13. Be skin test positive to seasonal and perennial aeroallergens that are present in the environment during the time that the subject is enrolled in the study, or if skin test positive to these aeroallergens the subject must not report worsening of symptoms when exposed to these aeroallergens during the time that the subject is participating in the study
14. Have a medical condition that in the opinion of the Investigator would impair the ability of the subject to participate
15. Have an inability to perform spirometry of acceptable quality
16. Be intolerant to Aridol, methacholine or albuterol
17. Be pregnant or lactating
18. Have participated in any other investigative drug study parallel to, or within 4 weeks of study entry
19. Be an Investigator, site employee or otherwise be directly affiliated with the study site including being a member of the immediate family of an Investigator, site employee (where an immediate family member is defined as spouse, parent, child or sibling, whether biological or legally adopted or in foster care)
20. Have a body mass index (BMI) ≥ 30
21. Have been diagnosed at Screening Visit (Visit 1) as definitively having or not having asthma; patients that will not continue in the study include those given the following diagnosis: asthma is extremely likely or definite (95 to 100% likelihood) or asthma is very unlikely or excluded (0 to < 5% likelihood)
22. Have previously been enrolled in this study at this or at any other clinical trials site
23. Have previously received an Aridol challenge
24. Have a clinically significantly abnormal chest x-ray

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240
Dates: Start 2005-11; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Comparison of Aridol and exercise BHR tests
Safety of Aridol test

SECONDARY OUTCOMES:
Comparison of Aridol and methacholine test
Comparison of Aridol test and clinical diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: David Pearlman, MD, Principal Investigator — Colorado Asthma and Allergy Centers, Denver, CO
Locations (1):
- Colorado Asthma and Allergy Centers, 125 Rampart Way, Denver, Colorado, United States

REFERENCES:
- [Background] Anderson SD, Brannan J, Spring J, Spalding N, Rodwell LT, Chan K, Gonda I, Walsh A, Clark AR. A new method for bronchial-provocation testing in asthmatic subjects using a dry powder of mannitol. Am J Respir Crit Care Med. 1997 Sep;156(3 Pt 1):758-65. doi: 10.1164/ajrccm.156.3.9701113. PMID 9309990
- [Background] Subbarao P, Brannan JD, Ho B, Anderson SD, Chan HK, Coates AL. Inhaled mannitol identifies methacholine-responsive children with active asthma. Pediatr Pulmonol. 2000 Apr;29(4):291-8. doi: 10.1002/(sici)1099-0496(200004)29:43.0.co;2-a. PMID 10738017
- [Background] Holzer K, Anderson SD, Chan HK, Douglass J. Mannitol as a challenge test to identify exercise-induced bronchoconstriction in elite athletes. Am J Respir Crit Care Med. 2003 Feb 15;167(4):534-7. doi: 10.1164/rccm.200208-916OC. Epub 2002 Nov 27. PMID 12456381
- [Background] Koskela HO, Hyvarinen L, Brannan JD, Chan HK, Anderson SD. Sensitivity and validity of three bronchial provocation tests to demonstrate the effect of inhaled corticosteroids in asthma. Chest. 2003 Oct;124(4):1341-9. doi: 10.1378/chest.124.4.1341. PMID 14555564